CLINICAL TRIAL: NCT02969200
Title: Fabry Disease: Renal Function During Long-term Enzyme Replacement Therapy Evaluated by Gold Standard GFR 51Cr-EDTA Clearance
Brief Title: Fabry: Renal Function During Long-term ERT by 51Cr-EDTA Clearance
Status: Completed | Type: Observational
Sponsor: Ulla Feldt-Rasmussen (Other)
Responsible Party: Sponsor-Investigator, Ulla Feldt-Rasmussen, Professor, Chief physician, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: FAB-KIDNEY
Record Dates: First submitted 2016-11-02; First posted 2016-11-21 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Fabry Disease
Keywords: Fabry Disease; Nephropathy; Measured GFR; Enzyme replacement therapy
MeSH Terms: conditions — Fabry Disease; Kidney Diseases | interventions — Enzyme Replacement Therapy; agalsidase beta; agalsidase alfa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Enzyme replacement therapy — All patients included in the study have received enzyme replacement therapy with either agalsidase alfa and/or agalsidase beta
  Other Names: Fabrazyme (agalsidase beta); Replagal (agalsidase alfa)

SUMMARY:
The aim of this study was to investigate renal function decline by measured glomerular filtration rate (mGFR) in patients with FD during enzyme replacement therapy, and to explore the influence of age on renal function in FD.

DETAILED DESCRIPTION:
Nephropathy is common in Fabry disease (FD). Renal function decline is often the first sign of major organ involvement, sometimes progressing to end-stage renal failure. Available studies of renal function during enzyme replacement therapy have shown inconsistent results, and are based on different composition of patient materials and follow-up time.

Most investigations have used estimated glomerular filtration rate (eGFR) for evaluating renal function. GFR is an important indicator of renal function. eGFR based on a serum creatinine measurement is most commonly used in FD. However, this method has been shown to be unreliable, as serum creatinine levels are influenced by other factors than renal function such as ethnic group, muscle mass, age, hydration and diet. Performance of eGFR in detecting minor changes in renal function is poor. A 10 year old review on renal function evaluation in patients with FD recommended the use of GFR based on an exogenous marker, e.g. Cr-EDTA. Nevertheless, only few studies have used mGFR for evaluation of renal function and to our knowledge, the present study is the first to describe the rate of renal function decline with consecutive mGFR values in a nationwide population of patients with FD.

Renal function declines with age in renal healthy individuals. To our knowledge, the present study is the first to age-standardize renal function in patients with FD to adjust for age-dependent renal deterioration.

ELIGIBILITY:
Inclusion Criteria:

* Genetically and/or enzymatically verified Fabry disease

Exclusion Criteria:

* End-stage renal disease prior to baseline (GFR <15 ml/min/1.73m2, dialysis or renal transplant)
* Patient has not received enzyme replacement therapy during follow-up
* Patient has had less than 3 measurement of GFR during follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Fabry disease
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2015-04; Primary Completion 2016-09 (Actual); Study Completion 2016-12-09 (Actual)

PRIMARY OUTCOMES:
measured glomerular filtration rate | Assessed every 6-12 months; from baseline and up to 15 years
  GFR was measured at least once a year by the one sample 51Cr-ethylenendiaminetetra acetic acid (EDTA) clearance technique using two (for duplicate determination) plasma samples 200 min after the injection of 4 (3.8-4.2) MBq 51Cr-EDTA. In children (< 15y) the injected 51Cr-activity was 3 MBq, and the blood-samples were collected 120 min after radiotracer injection. (< 5y: 2 MBq).

SECONDARY OUTCOMES:
urinary protein excretion | Assessed every 6-12 months; from baseline and up to 15 years
  Repeated twenty-four hour urine samples were collected by patients at home, the last 24 hours before coming to the hospital. These samples were analysed for albumin, creatinine and protein. Furthermore spot urine samples were applied and analysed for albumin, creatinine and protein. Albumin-creatinine-ratio was calculated and abnormal values were defined as > 30 mg/g. Urine protein- and albumin values below detection limit (< 0.04 g/L and < 3 mg/L, respectively) were converted to zero for statistical analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Ulla V Feldt-Rasmussen, MD, DMSc, Principal Investigator — Department of Medical Endocrinology, Copenhagen University Hospital, Rigshospitalet
Locations (1):
- National University Hospital, Department of Medical Endocrinology, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No